CLINICAL TRIAL: NCT06734416
Title: Evaluation of the Role of Brain Natriuretic Peptide in Acute Coronary Syndrome .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Gamal kamel Mohamed, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: BNP IN ACS
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndromes
Keywords: Brain natriuretic peptide
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: patients with Acute Coronary Syndrome , this group will be sub classified into: Non-ST-elevation myocardial infarction (NSTEMI) ST-elevation myocardial infarction (STEMI) Unstable angina
- group 2: apparently healthy patients will be included in this study as a control group for comparison

SUMMARY:
The measurements of the natriuretic peptide are useful and beneficial for risk stratification irrespective of the cause during admission time or during hospital stay course. the aim of the study is to Assessment of the role of Brain natriuretic peptide in diagnosis of acute coronary syndrome . Evaluation of the relation of Brain natriuretic peptide to the severity and occurrence of complications in acute coronary syndrome .

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) is regarded as one of the important leading causes of disability and death across the globe.

Acute coronary syndrome (ACS) applies to a variety of events reporting ischemia, ranging from stable angina without myocardial necrosis to ST -segment elevation myocardial infarction (STEMI). The need for prevention and detection of coronary vascular disease as early as possible by using newer and more cost effective tools is suggested . For risk stratification in patients with ACS, serial ECG monitoring and cardiac biomarkers measurement are needed as part of the diagnostic workup. B-type natriuretic peptide is synthesized as a high molecular weight precursor pro-brain natriuretic peptide (BNP) which is cleaved to release BNP and the amino-terminal fragment, N-terminal pro (NT-pro) BNP. Both peptides are released from the cardiac ventricles in response to the increased wall stress and hence its levels may indicate ventricular strain BNP is believed to have its role as natriuretic hormone and vasodilation. Among other effects are inhibition of the Renin Angiotensin-Aldosterone system(RAAS), and sympathetic nervous system. After an ischemic occurrence, BNP levels peak in 14 to 40 hours .

ELIGIBILITY:
Inclusion Criteria:

* patients with acute coronary syndrome.

Exclusion Criteria:

* Patients with previous MI
* Eection fraction (EF) less than 30%
* Patients having cardiomyopathy
* Patients having renal, liver, malignant, infectious, or inflammatory diseases .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Brain natriuretic peptide level in blood | baseline
  level of Brain natriuretic peptide in acute coronary syndrome patients.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volterrani M, Iellamo F, Senni M, Piepoli MF. Therapeutic options of Angiotensin Receptor Neprilysin inhibitors (ARNis) in chronic heart failure with reduced ejection fraction: Beyond RAAS and sympathetic nervous system inhibition. Int J Cardiol. 2017 Jan 1;226:132-135. doi: 10.1016/j.ijcard.2016.04.180. Epub 2016 May 7. PMID 27184730
- [Background] Mukoyama M, Nakao K, Hosoda K, Suga S, Saito Y, Ogawa Y, Shirakami G, Jougasaki M, Obata K, Yasue H, et al. Brain natriuretic peptide as a novel cardiac hormone in humans. Evidence for an exquisite dual natriuretic peptide system, atrial natriuretic peptide and brain natriuretic peptide. J Clin Invest. 1991 Apr;87(4):1402-12. doi: 10.1172/JCI115146. PMID 1849149